CLINICAL TRIAL: NCT00252044
Title: The Dopaminergic System in Schizotypal Personality Disorder: Pergolide for Cognitive Symptoms in Schizotypal Personality Disorder
Brief Title: Pergolide for Cognitive Symptoms in Schizotypal Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 7609-028
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2005-11-21 (Estimated); Status verified 2005-11

CONDITIONS: Schizotypal Personality Disorder; Other Personality Disorders
MeSH Terms: conditions — Schizotypal Personality Disorder | interventions — Pergolide

INTERVENTIONS:
Drug: Pergolide

SUMMARY:
Hypothesis: Schizotypal personality disorder patients will show cognitive improvements in 1) working memory 2) learning and memory 3) sustained attention 4) enhanced performance on the AX-CPT, N-back and Eriksen during pergolide treatment. There will be a significant diagnosis by drug administration of 0.3 mg of oral pergolide interaction for performance on the cognitive tasks, with the schizotypal personality disorder group demonstrating significantly improved peformance compared to the other personality disorder group after pergolide compared with placebo.

Design: Randomized, double-blind, crossover study of pergolide vs. placebo. Half of subjects receive pergolide for eight weeks; half of subjects receive placebo for four weeks followed by pergolide for four weeks.

ELIGIBILITY:
Inclusion Criteria: DSM-IV criteria for Schizotypal Personality Disorder (or meets full criteria bar one) or another personality disorder and shows impairment on markers of cognitive functioning. Medically healthy, not abusing drugs or alcohol, is at least two weeks medication-free and does not have significant neurological disease.

-

Exclusion Criteria: DSM-IV or RDC criteria for Schizophrenia or any Schizophrenia-related psychotic disorder or for Bipolar Disorder. Any other Axis I disorders must be transient and preceded by the personality disorder diagnosis, which should be primarily responsible for subject's functional impairment.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2000-10

PRIMARY OUTCOMES:
Performance on tests of sustained attention, episodic memory and working memory at baseline and after 2, 4, 6 and 8 weeks on the study medication

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale, Positive and Negative Symptom Scale and Clinical Global Impression scale at baseline and then weekly through the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Siever, MD, Principal Investigator — Bronx VA Medical Center/Mount Sinai School of Medicine
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States